CLINICAL TRIAL: NCT06448533
Title: The Predictive Value of Prostate Spherical Volume Ratio in Lower Urinary Tract Symptoms and Clinical Progression of Benign Prostatic Hyperplasia:A Single-center Paired Validating Confirmatory Study
Status: Completed | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1.0 2022.9.10
Record Dates: First submitted 2024-06-02; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Lower Urinary Tract Symptoms，Prostatic Hyperplasia
Keywords: Lower Urinary Tract Symptoms，prostatic hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study was a retrospective cohort study clinical trial designed to assess the predictive ability of the prostate morphometric parameter, Prostate Spherical Volume Ratio, in the lower urinary tract symptoms and clinical progression of benign prostatic hyperplasia; and to compare the predictive ability of other anatomical parameters of the prostate (prostatic urethral length, intravesical prostatic protrusion, presumed circle area ratio, and prostate volume) in the lower urinary tract symptoms and clinical progression of benign prostatic hyperplasia

DETAILED DESCRIPTION:
This was a retrospective observational study approved by the Ethics Committee of Shanghai Oriental Hospital. We collected patients with BPH who underwent MRI, urine flow measurement and completed the IPSS questionnaire in our hospital between September 2022 and April 2023, measured each anatomical parameter of the patient's prostate by MRI, analysed the relationship of these prostate parameters with IPSS and urine flow, and conducted a follow-up of the clinical progression of the prostate in these patients to evaluate the predictive efficacy of prostate parameters for LUTS and clinical progression of benign prostatic hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* All patients had obvious lower urinary tract symptoms such as urinary frequency, increased nocturia, and a feeling of incomplete urination, etc. They all completed prostate MRI, IPSS questionnaire, and uroflowmetry for a clear diagnosis of BPH.

Exclusion Criteria:

* 1, previous history of bladder, prostate, urethra surgery; 2, the existence of other diseases that cause urinary dysfunction: such as neurogenic bladder, bladder stones, urethral stenosis, urinary tract infections, acute prostatitis, etc.; 3, the existence of mental, mental disorders, can not be accurately expressed and family members can not help to improve the IPSS scores; 4, to receive prostatic hyperplasia medication, such as: α-blocker therapy, 5α reductase inhibitors, etc. have not been discontinued for 6 months; 5, refused to participate in this study

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male with benign prostatic hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
clinical progression of benign prostatic hyperplasia | 1 year of observation and follow-up after enrolment
  The primary outcome, described as clinical progression of benign prostatic hyperplasia, was the first occurrence of an increase in the IPSS of at least 4 points, benign prostatic hyperplasia-related prostatic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji T, Huang K, He B, Wang H. The predictive value of prostate spherical volume ratio in lower urinary tract symptoms and clinical progression of benign prostatic hyperplasia: a retrospective cohort study. Int Urol Nephrol. 2025 Jul;57(7):2023-2032. doi: 10.1007/s11255-024-04355-4. Epub 2025 Jan 15. PMID 39812965